CLINICAL TRIAL: NCT07146490
Title: Effects of Exercise Intensity on Neurochemical and Cognitive Function: The Role of Lactate and Irisin
Brief Title: Effects of Different Types of Exercise on Irisin and Cognitive Performance (Exercise-Irisin)
Acronym: Ex-Irisin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aksaray University Training and Research Hospital (Other)
Responsible Party: Principal Investigator, serkan pancar, Assoc. Prof., Aksaray University Training and Research Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 10.03
Record Dates: First submitted 2025-08-20; First posted 2025-08-28 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Irisin; Lactate; Cognitive Function; Exercise Training
Keywords: HIIT; Irisin; Lactate; Cognitive Function

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low-Intensity Continuous Training Group (n=4) (Experimental): They were asked to perform low intensity exercise for the specified time, determined according to their maximal oxygen consumption capacity.
  Interventions: Behavioral: Low Exercise
- Long-interval high-Intensity Interval Training Group (n=4) (Experimental): They were asked to perform long interval moderate intensity exercise for the specified time, determined according to their maximal oxygen consumption capacity.
  Interventions: Behavioral: Long Interval Exercise
- Short-interval high-Intensity Interval Training Group (n=4) (Experimental): They were asked to perform short interval high intensity exercise for the specified time, determined according to their maximal oxygen consumption capacity.
  Interventions: Behavioral: Short Intevral Exercise

INTERVENTIONS:
Behavioral: Low Exercise — Low-Intensity Continuous Training (LICT): Participants ran continuously for 24 minutes at 50-60% of their MAS without breaks.
  Arms: Low-Intensity Continuous Training Group (n=4)
Behavioral: Long Interval Exercise — Long-interval high-Intensity Interval Training (LI-HIIT): Participants ran at a speed corresponding to 80-90% of their MAS. The protocol consisted of four 4-minute bouts, separated by 2-minute active recovery periods, during which participants ran at 50% of their MAS. This pattern totaled 24 minutes of exercise.
  Arms: Long-interval high-Intensity Interval Training Group (n=4)
Behavioral: Short Intevral Exercise — Short-interval high-Intensity Interval Training (SI-HIIT): Participants ran at 110-120% of their MAS for 15-second intervals, covering a pre-calculated distance during each bout. After each 15-second sprint, they rested passively for 15 seconds and returned to their starting point. This was repeated continuously for 3 minutes, constituting one set. A total of four 3-minute sets were completed, interspersed with 3-minute passive rest periods, yielding a total exercise time of 24 minutes.
  Arms: Short-interval high-Intensity Interval Training Group (n=4)

SUMMARY:
Purpose The purpose of this study was to determine the acute effects of different exercise intensities on Irisin levels, trail making test performance, and feeling scale.

Method

This randomized crossover controlled trial aims to examine the acute effects of three experimental conditions-Short-Interval High-Intensity Interval Training (SI-HIIT), Long-Interval High-Intensity Interval Training (LI-HIIT) and Low-Intensity Continuous Training (LICT), on cognitive performance (via the Trial Making Test, ) and associated neurochemical responses (e.g., serum Irisin and blood lactate levels) in healthy young adults aged 18-25 years.

All participants completed the three conditions in a randomized and counterbalanced manner. To ensure balanced exposure, they were assigned to one of three groups (n = 4 per group), each following a distinct condition order based on a Latin square design. This approach guaranteed that each session occurred equally across time points (sessions 1-3) and that the order minimized sequence effects by rotating the position of each condition relative to the others.

To control for potential carryover-particularly from elevated neurochemical responses following intense exercise (Irisin increases reported -no two high-intensity sessions were scheduled consecutively. Where possible, higher and lower intensity protocols were be alternated. Furthermore, a seven-day interval separated each session to reduce residual physiological or cognitive effects.

The trial protocol was developed in line with CONSORT and SPIRIT guidelines, including relevant extensions for within-subject designs and non-pharmacological interventions. Participants were blinded to the study hypothesis.

All exercise sessions conducted under supervision of a certified strength and conditioning coach to ensure consistency and adherence to protocol in the morning (09:00-11:00) on a track and field pitch to control for chronobiological variation. Participants were instructed to avoid strenuous activity for 48 hours prior, abstain from alcohol and caffeine for 24 hours, and obtain at least 7-8 hours of sleep before each session. Dietary habits and general lifestyle were to remain unchanged throughout the study.

During the first visit, participants' body weight and body fat percentage were assessed using bioelectrical impedance analysis. Resting heart rate was then recorded, followed by administration of the Yo-Yo Intermittent Recovery Test Level 1 to determine maximal aerobic speed, aerobic capacity, and peak heart rate.

In the following four visits, each participant completed all experimental conditions. Each exercise session began with a standardized 10-minute warm-up, including light jogging, dynamic stretching, and movement preparation drills.

All exercise sessions were conducted on a standard track and field facility and lasted 40 minutes in total, consisting of a 10-minute standardized warm-up, 24 minutes of exercise, and a 5-minute recovery period. The exercise component was individually prescribed based on each participant's maximal aerobic speed, determined from the Yo-Yo Intermittent Recovery Test Level 1. All running distances were calculated individually using time × speed formulas based on each participant's maximal aerobic speed, ensuring workload equivalence across conditions.

* Short-interval high-Intensity Interval Training: Participants ran at 110-120% of their MAS for 15-second intervals.
* Long-interval high-Intensity Interval Training: Participants ran at a speed corresponding to 80-90% of their MAS.
* Low-Intensity Continuous Training: Participants ran continuously for 24 minutes at 50-60% of their MAS without breaks.

Venous blood samples were collected before and immediately after each session to assess neurochemical markers. Subsequently, cognitive performance was evaluated using the computerized Trial Making Test to measure executive function. Heart rate was continuously monitored during all exercise conditions using a Polar V800 device. Following each session, psychophysiological responses were assessed using the Feeling Scale.

ELIGIBILITY:
Inclusion Criteria

* Aged between 18 and 25 years
* No known medical condition that prevents participation in exercise
* Not currently using any pharmacological agents

Exclusion Criteria:

* Experiencing any discomfort before, during, or after exercise
* Current or past diagnosis of pharmacological or doping substance use
* Engaging in regular exercise (more than 3 times per week) within the last 2 weeks
* History of alcohol or substance addiction
* Any other condition or factor that may prevent full participation in the study protocol

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Only male participants are eligible to participate in this study based on biological sex.
Enrollment: 12 (Actual)
Dates: Start 2025-06-10 (Actual); Primary Completion 2025-07-27 (Actual); Study Completion 2025-08-05 (Actual)

PRIMARY OUTCOMES:
Lactate | Baseline and immediately after exercise (Day 1)
  Lactate levels were measured in millimoles per liter (mmol/L) from capillary/venous blood samples taken before and after exercise using a lactate analyzer.
Irisin | Baseline and immediately after exercise (Day 1)
  Irisin levels were measured using a Sunred brand ELISA kit from blood samples taken baseline and after exercise, and the results were reported in pg/mL units.
Trial Making Test | Baseline and immediately after exercise (Day 1)
  The Trail Making Test (TMT) is a widely used neuropsychological assessment tool to evaluate attention, visual scanning, processing speed, mental flexibility, and executive function.
  TMT-A measures processing speed and visual attention by requiring participants to connect sequential numbers (1-25) as quickly as possible. Completion times were recorded in seconds.
  TMT-B measures cognitive flexibility and executive control by requiring participants to alternate between numbers and letters (1-A-2-B, etc.).
Feeling Scale | Baseline and immediately after exercise (Day 1)
  The Feeling Scale (FS) is a single-item measure of affective valence during or after exercise. Participants are asked, "How are you feeling right now?" and respond on an 11-point bipolar scale ranging from -5 to +5.
  Scoring:
  -5 = Very Bad
  0 = Neutral
  +5 = Very Good
  Negative scores indicate unpleasant affect, whereas positive scores indicate pleasant affect. Higher scores reflect better subjective feelings.

CONTACTS AND LOCATIONS:
Overall Officials: serkan PANCAR, Assistant Professor, Study Director — Aksaray University /Faculty of Sports Sciences
Locations (1):
- Aksaray University, Aksaray, Center, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided